CLINICAL TRIAL: NCT03437473
Title: A Randomized Controlled Study of the Safety and Efficacy of Neurostimulation Using a Vagus Nerve Stimulation Device in Patients With Rheumatoid Arthritis
Brief Title: Safety and Efficacy of Vagus Nerve Stimulator in Patients With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SetPoint Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: SPM-008
Record Dates: First submitted 2018-02-06; First posted 2018-02-19 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Active stimulation QD (Active Comparator)
  Interventions: Device: SetPoint Medical Neurostimulation of the Cholinergic Anti-inflammatory Pathway System
- Active stimulation QID (Active Comparator)
  Interventions: Device: SetPoint Medical Neurostimulation of the Cholinergic Anti-inflammatory Pathway System
- No stimulation (Sham Comparator)
  Interventions: Device: SetPoint Medical Neurostimulation of the Cholinergic Anti-inflammatory Pathway System

INTERVENTIONS:
Device: SetPoint Medical Neurostimulation of the Cholinergic Anti-inflammatory Pathway System — Active Implantable Vagus Nerve Stimulation device.
  Other Names: SetPoint System

SUMMARY:
Multi-site, first-in-human study to assess safety and efficacy of an active implantable Vagus Nerve Stimulation (VNS) device in 15 adult patients with active moderate-to-severe rheumatoid arthritis who have had an incomplete response or intolerability to at least two different mechanisms of action.

DETAILED DESCRIPTION:
This is a two-stage study where Stage 1 is open label, and Stage 2 is randomized and sham controlled where the sites and subjects are blinded to treatment. Three subjects will be enrolled in Stage 1 of the study. And 12 subjects will be enrolled in Stage 2. Subjects will be treated for a total of 12 weeks.

Subjects will be asked to visit the clinic at day 0, week 1-6, week 8 and week 12. During these visits, the following activities will be conducted: standard patient and physician assessments of RA activity, blood sample collection for RA biomarkers, and a hand MRI.

Subjects who complete the study will have the option to enroll in a long-term extension study. Subjects that do not participate in the extension study can opt to either have their device permanently inactivated and left in place or have the device surgically explanted.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female and 22-75 years of age, inclusive
2. Have provided informed consent
3. Have a diagnosis of adult-onset rheumatoid arthritis as defined by the 2010 ACR/EULAR classification criteria (Aletaha, 2010)
4. Have moderately to severely active RA defined by at least 4/28 tender and 4/28 swollen joints and CDAI score >10
5. Have been treated at approved doses with at least 2 biologic DMARDs and/or new targeted synthetic DMARDs (e.g. JAK inhibition) for at least 3 months and either:

   1. experienced insufficient efficacy or loss of efficacy
   2. experienced intolerance of such treatment
6. Have had regular use of at least 1 conventional DMARDs for at least the 12 weeks prior to study entry with a continuous, non-changing dose for at least 8 weeks prior to screening visit
7. Women of childbearing potential must not be pregnant at the time of screening and must agree to use a double barrier method of contraception throughout the study

Exclusion Criteria:

1. Have taken the following within the defined time period prior to screening visit:

   i. Rituximab: 6 months ii. Infliximab, golimumab, adalimumab, certolizumab pegol, tocilizumab: 60 days iii. Abatacept, etanercept, anakinra: 30 days iv. Tofacitinib: 30 days v. Investigational biologic agents: 6 months for depleting agents, 60 days for others vi. Investigational small molecules: 5 times the pharmacokinetic half-life or 30 days, whichever is longer vii. Intra-articular corticosteroid injection: 30 days
2. Are currently receiving corticosteroids at doses greater than 10 mg per day of prednisone (or equivalent) or have been receiving an unstable dosing regimen of corticosteroids within 2 weeks of screening visit
3. Have started treatment with non-steroidal anti-inflammatory drugs (NSAIDs) or have been receiving an unstable dosing regimen of NSAIDs within 2 weeks of screening visit
4. Documented significant psychiatric illness or substance abuse
5. Active infection requiring treatment with antibiotics
6. Uncontrolled hypertension
7. Uncontrolled diabetes
8. History of stroke
9. Known cardiac disease, including cardiomyopathy with ejection fraction <40%, recent myocardial infarction or unstable angina, or heart failure with New York Heart Association class III or IV symptoms
10. Known neurological syndromes
11. Known atherosclerotic disease including contralateral carotid artery
12. BMI <18.5 or >35
13. Any condition per the investigator's clinical judgment that precludes participation in the study

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
incidence of Adverse Events | Enrollment to Week 12
  treatment-emergent incidence rates of Adverse Events, Adverse Device Effects, Serious Adverse Events, Serious Adverse Device Effects, Unanticipated Adverse Device Effects, and Unanticipated Serious Adverse Device Effects

SECONDARY OUTCOMES:
change in Disease Activity Score (DAS) 28 - C-reactive protein (CRP) | change from baseline at Day 0 and Week 12
  comparison between the active device group and the inactive device group of the change in DAS28-CRP
change in American College of Rheumatology (ACR) 20, 50 and 70 response rates | change from baseline at Day 0 and Week 12
  comparison between the active device group and the inactive device group of the change in ACR 20/50/70
change in European League Against Rheumatism (EULAR) response and remission rate | change from baseline at Day 0 and Week 12
  comparison between the active device group and the inactive device group of the change in EULAR
change in hand MRI | change from baseline at Day 0 and Week 12
  comparison between the active device group and the inactive device group of the change in Outcomes Measures in Rheumatology Rheumatoid Arthritis MRI Scoring System (OMERACT RAMRIS) hand MRI index of synovitis

CONTACTS AND LOCATIONS:
Overall Officials: Mark Genovese, MD, Study Director — Stanford University
Locations (4):
- United States (4):
  - Arthritis & Rheumatic Disease Specialties, Aventura, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Northwell Health Division of Rheumatology, Great Neck, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Genovese MC, Gaylis NB, Sikes D, Kivitz A, Lewis Horowitz D, Peterfy C, Glass EV, Levine YA, Chernoff D. Safety and efficacy of neurostimulation with a miniaturised vagus nerve stimulation device in patients with multidrug-refractory rheumatoid arthritis: a two-stage multicentre, randomised pilot study. Lancet Rheumatol. 2020 Sep;2(9):e527-e538. doi: 10.1016/S2665-9913(20)30172-7. Epub 2020 Jul 28. PMID 38273617